CLINICAL TRIAL: NCT06890494
Title: Clinical Study on the Safety and Efficacy of BiTE-EV Therapy in Relapsed/Refractory Acute B-Cell Lymphoblastic Leukemia
Brief Title: Clinical Study on the Safety and Efficacy of BiTE-EV in Relapsed/Refractory Acute B-Cell Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-054
Record Dates: First submitted 2025-02-04; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BiTE-EV therapy (Experimental)
  Interventions: Drug: BiTE-EV

INTERVENTIONS:
Drug: BiTE-EV — Thi product organically combines extracellular vesicles with BiTEs, and enables stable expression of the bispecific antibody on the surface of mesenchymal stem cells. By collecting the culture supernatant, the bispecific vesicles BiTE-EV, which express both CD3 and CD19 antibodies on their surface, are enriched and isolated.

SUMMARY:
The goal of this clinical trial is to learn if BiTE-EV works to treat relapsed/refractory acute B-cell leukemia in adults. It will also learn about the safety of BiTE-EV. The main questions it aims to answer are:

Can BiTE-EV effectively treat relapsed/refractory acute B-cell lymphoblastic leukemia? What medical problems do participants have when taking BiTE-EV?

Participants will:

Take BiTE-EV every other day for 1 or 2 months Keep a diary of their symptoms during the medication period During the follow-up period, visit the clinic once every 4 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria: Patients can be enrolled in the group only if they meet all of the following conditions:

* Patients with acute B lymphocytic leukemia who are clinically diagnosed as relapsed (relapsed after CAR-T treatment or relapsed after transplantation), refractory, or whose T cells cannot be used for the production of CAR-T cells.
* Tumor cells show positive expression of CD19 detected by flow cytometry or immunohistochemistry.
* The age is between 18 and 70 years old (inclusive).
* The expected survival period from the date of signing the informed consent form is greater than 3 months.
* The Eastern Cooperative Oncology Group (ECOG) performance status score is ≤ 2.
* The functions of vital organs should meet the following requirements:

  * The ejection fraction (EF) is > 50%, and there is no significant abnormality in the electrocardiogram.
  * The peripheral oxygen saturation (SpO2) is ≥ 92%.
  * The serum creatinine (Cr) is ≤ 1.5 times the upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are ≤ 5 times the upper limit of normal (ULN), and total bilirubin (TBil) is ≤ 3 times the upper limit of normal (ULN).
* Subjects with pregnancy plans must agree to take contraceptive measures before enrolling in the study and six months after the study. If the subject is pregnant or suspected to be pregnant, they should immediately notify the investigator.
* The subject or the guardian understands and signs the informed consent form.

Exclusion Criteria:If any one of the following conditions is met, the subject cannot be enrolled in the group:

* Complicated with other diseases that are not effectively controlled, including but not limited to persistent or poorly controlled infections, symptomatic congestive heart failure, unstable angina pectoris, arrhythmia, poorly controlled pulmonary diseases or mental disorders.
* Having other active malignant tumors.
* Complicated with severe infections that cannot be effectively controlled.
* Those who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), and those with peripheral blood hepatitis B virus (HBV) DNA higher than the detection limit need to be excluded; those who are positive for hepatitis C virus (HCV) antibody and positive for peripheral blood HCV RNA need to be excluded; those with positive cytomegalovirus (CMV) DNA detection; those with positive peripheral blood Epstein-Barr virus (EBV) DNA detection.
* Those who are positive for human immunodeficiency virus (HIV) antibody test or positive for syphilis test.
* Having a history of severe allergy to biological products (including antibiotics).

Patients with relapsed after allogeneic hematopoietic stem cell transplantation who have experienced grade 3 - 4 acute graft-versus-host disease (GvHD).

* Female subjects who are pregnant or in the lactation period.
* Active autoimmune diseases that require systemic immunosuppressive treatment.
* Situations that the investigator believes may increase the risk of the subject or interfere with the test results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events (TRAEs) | 3 months
  The number of participants experiencing treatment-related adverse events during the study.
  Assessment: Number of participants with at least one TRAE. Unit of Measure: Number of participants
Severity of Treatment-Related Adverse Events | 3 months
  The severity of TRAEs, graded according to CTCAE version X. Assessment: Maximum CTCAE grade for each TRAE per participant. Unit of Measure: CTCAE grade (1, 2, 3, 4, or 5)
Frequency of Treatment-Related Adverse Events | 3 months
  The number of occurrences of each specific TRAE during the study. Assessment: Number of events for each specific TRAE. Unit of Measure: Number of events
Type of Treatment-Related Adverse Events | 3 months
  The specific types of TRAEs observed during the study. Assessment: List of all TRAEs observed, classified by system organ class and preferred term according to MedDRA (or other standard medical dictionary).
  Unit of Measure: Categorical (System Organ Class and Preferred Term)

SECONDARY OUTCOMES:
the efficacy of BiTE-EV in the treatment of relapsed/refractory acute B-cell lymphoblastic leukemia. | 2 years
  Outcome Measure 1: Treatment response assessed at the end of the first and second treatment cycles. Assessment: Complete Remission (CR)，CR with incomplete hematologic recovery (CRi)，Partial Remission (PR)，No Response (NR)，Stable Disease (SD)，Progressive Disease (PD)，Unit of Measure: Categorical (CR, CRi, PR, NR, SD, PD) Outcome Measure 2: Quantitative assessment of MRD clearance in fusion gene-positive leukemia patients.Assessment: MRD Level，Unit of Measure: e.g., log10 reduction, MRD positive/negative, or % MRD (specify actual unit) Outcome Measure 3: Duration of response in patients who complete treatment without further anti-leukemic therapy.Assessment: Time from initial response to relapse or progression.Unit of Measure: Months Outcome Measure 4: Leukemia-free survival in patients who complete treatment without further anti-leukemic therapy.Assessment: Time from initial response to relapse or death from leukemia-related causes.Unit of Measure: Months
Maximum Concentration (Cmax) | 2 months
  The maximum concentration of BiTE-EV accumulated in peripheral blood during infusion.
  Assessment: Maximum concentration Unit of Measure: ng/mL
Time to Maximum Concentration (Tmax) | 2 months
  The time to reach the maximum concentration of BiTE-EV in peripheral blood during infusion.
  Assessment: Time to maximum concentration Unit of Measure: hours (h)
Half-life (t½) | 2 months
  The half-life of BiTE-EV in peripheral blood. Assessment: Half-life Unit of Measure: hours (h)
Area Under the Curve (AUC28d) | 28 days
  The 28-day area under the plasma concentration versus time curve for BiTE-EV. Assessment: Area under the curve from time 0 to 28 days. Unit of Measure: ng*h/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, China